CLINICAL TRIAL: NCT06129851
Title: Quantifying Optimal Relugolix Duration With Radiation in High Risk Prostate Cancer (QURE-PC)
Brief Title: Relugolix in Combination With Radiation Therapy for Treating Patients With High Risk Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Xinglei Shen, Principal Investigator, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150674; NCI-2023-09079 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00150674 (Other: University of Kansas Cancer Center); P30CA168524 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Brachytherapy; Absorptiometry, Photon; Bone Density; Congresses as Topic; Radiation; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (relugolix, brachytherapy, external beam radiation) (Experimental): Patients receive relugolix PO QD. Cycles repeat every 3 months for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 30 to 180 days after start of relugolix, patients undergo brachytherapy and external beam radiation over 25 fractions. Patients undergo bone scan, CT or MRI or PSMA PET scan during screening. Patients also undergo DEXA scan and may optionally undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Radiation: Brachytherapy; Procedure: Computed Tomography; Procedure: Dual X-ray Absorptiometry; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Other: Questionnaire Administration; Drug: Relugolix
- Arm B (relugolix, brachytherapy, external beam radiation) (Experimental): Patients receive relugolix PO QD. Cycles repeat every 3 months for 24 months in the absence of disease progression or unacceptable toxicity. Beginning 30 to 180 days after start of relugolix, patients undergo brachytherapy and external beam radiation over 25 fractions. Patients undergo bone scan, CT or MRI or PSMA PET scan during screening. Patients also undergo DEXA scan and may optionally undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Radiation: Brachytherapy; Procedure: Computed Tomography; Procedure: Dual X-ray Absorptiometry; Radiation: External Beam Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Other: Questionnaire Administration; Drug: Relugolix

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Radiation: Brachytherapy — Undergo brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Dual X-ray Absorptiometry — Undergo DEXA scan
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA (Bone Density); DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: PSMA PET Scan — Undergo PSMA PET
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Other: Questionnaire Administration — Ancillary studies
Drug: Relugolix — Given PO
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385

SUMMARY:
This phase II trial evaluates the best duration for relugolix to be given in combination with radiation therapy when treating patients with high risk prostate cancer. Prostate cancer is a hormonal influenced cancer. Part of the usual treatment for patients with prostate cancer is androgen deprivation therapy (ADT). ADT is used to lower the amount of testosterone in the body, because testosterone appears to help prostate cancer grow. Relugolix works to reduce testosterone levels, which may inhibit proliferation of prostate cancer cells. It is approved by the Food and Drug Administration to treat prostate cancer. Adding relugolix to standard radiation therapy might work better and have fewer side effects than prior forms of hormonal therapy, but the optimal duration of relugolix in combination with radiation is not known.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the biochemical recurrence rate between 12 and 24 months of relugolix in patients with high risk prostate cancer treated with combination external beam radiation and brachytherapy.

SECONDARY OBJECTIVES:

I. To compare the composite quality of life in patient treated with 12 months and 24 months of relugolix as assessed by the Expanded Prostate Composite Index Short Form (EPIC-26) instrument.

II. To compare the treatment related toxicity between 12 months and 24 months of relugolix as assessed by Common Terminology Criteria for Adverse Events version 5.0. (CTCAE v 5.0) criteria.

III. To compare the rate of major adverse cardiovascular events (MACE) in patients treated with 12 and 24 months of relugolix.

IV. To establish the rate of patient compliance using patient reported drug diary.

V. To compare the rate of testosterone recovery after 12 and 24 months of relugolix.

EXPLORATORY OBJECTIVE:

I. To establish Decipher genomic classifier as predictor of cancer control.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive relugolix orally (PO) once daily (QD). Cycles repeat every 3 months for 12 months in the absence of disease progression or unacceptable toxicity. Beginning 30 to 180 days after start of relugolix, patients undergo brachytherapy and external beam radiation over 25 fractions. Patients undergo bone scan, computed tomography (CT) or magnetic resonance imaging (MRI) or prostate-specific membrane antigen (PSMA) positron emission tomography (PET) scan during screening. Patients also undergo dual x-ray absorptiometry (DEXA) scan and may optionally undergo blood sample collection throughout the trial.

ARM B: Patients receive relugolix PO QD. Cycles repeat every 3 months for 24 months in the absence of disease progression or unacceptable toxicity. Beginning 30 to 180 days after start of relugolix, patients undergo brachytherapy and external beam radiation over 25 fractions. Patients undergo bone scan, CT or MRI or PSMA PET scan during screening. Patients also undergo DEXA scan and may optionally undergo blood sample collection throughout the trial.

After completion of study treatment, patients in Arm A are followed up every 3 months for 12 months and then every 6 months for up to 36 months and patients in Arm B are followed up every 6 months for up 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant or Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Life expectancy > 5 years
* Patient diagnosed with National Comprehensive Cancer Network (NCCN) high risk and very high risk prostate cancer.

  * High risk is defined as:

    * T3a or
    * Grade group 4 or 5 or
    * Prostate-specific antigen (PSA) > 20 ng/mL
  * Very high risk is defined as:

    * T3b to T4 or
    * Primary Gleason pattern 5 or
    * Two or three high-risk features or
    * > 4 cores with grade group 4 or 5
* Eligible for treatment with combination brachytherapy, external beam radiation, and ADT
* Leukocytes >= 1.0 K/UL
* Platelets >= 100 K/UL
* Hemoglobin ≥ 9 g/dL
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal (ULN)
* Men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed for the duration of study participation and for 2 weeks following completion of relugolix therapy

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Has a known allergic reaction to any excipient or component contained in the study drug formulation
* Active grade 3 (per the National Cancer Institute [NCI] CTCAE, version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment
* Current androgen deprivation therapy (unless testosterone > 50 ng/dL). Please note prior or concurrent bicalutamide at 50 mg/daily or less is allowed. Prior androgen deprivation therapy is allowed if testosterone has recovered to > 50 ng/dL
* Prolonged echocardiogram corrected QT (QTc) interval > 440 ns
* Prior pelvic therapy that would significantly overlap with radiation treatment fields
* Prior prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2025-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence | Up to 3 years
  Will be defined as serum prostate-specific antigen (PSA) level of nadir + 2 ng/mL by blood test.

SECONDARY OUTCOMES:
Composite quality of Life | Up to 5 years
  Will be assessed by the Expanded Prostate Composite Index Short Form (EPIC-26) and will be compared between the 2 arms in terms of hormonal domain and sexual domain of EPIC-26. An area under the curve (AUC) metric will be utilized to account for the overall quality of life from baseline through 36 months for each patient. A mixed effect model will be employed to construct an estimate of the difference in AUC between Arms A and B, including fixed effects of time, arm, and baseline characteristics (two or three covariates depending on the available sample size). A two-sample t-test with a significance level of 0.05 will be performed.
Incidence of adverse events | Up to 5 years
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0 and will be reported descriptively.
Incidence of major adverse cardiovascular events | Up to 5 years
  Will be assessed by medical record review and will be reported descriptively.
Participant compliance | Up to 2 years
  Will be assessed by patient study diary.
Time to testosterone recovery | Up to 5 years
  Will be assessed by blood tests and the percentage of patients in each arm who achieved baseline level or minimum 280 ng/dL will be reported at 3-month intervals up through 36 months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Xinglei Shen, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States